CLINICAL TRIAL: NCT06599658
Title: The Immunogenicity and Safety of COVID-19 and Influenza Vaccine Co-administration and Interval in Immunocompromised Hosts
Brief Title: COVID-19 Booster and IIV Schedule in Immunocompromised Hosts
Acronym: CO2I2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Ruth Sapir-Pichhadze, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2025-10781
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: COVID 19; Influenza; Rheumatoid Arthritis (RA); Systemic Lupus Erthematosus; Inflammatory Bowel Disease; Solid Organ Transplant Recipients; Immunocompromised Host; People Living With HIV
Keywords: Vaccine; Immunogenicity; Safety
MeSH Terms: conditions — COVID-19; Influenza, Human; Arthritis, Rheumatoid; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1 (Experimental): Covid-19 booster every 3 months and Inactivated influenza vaccine (IIV) at baseline
  Interventions: Biological: Inactivated influenza vaccine (IIV) at baseline; Biological: COVID-19 Vaccines at a 3-month interval
- Group 2 (Experimental): Covid-19 booster every 3 months and IIV at 1 month
  Interventions: Biological: COVID-19 Vaccines at a 3-month interval; Biological: Inactivated influenza vaccine at Month 1
- Group 3 (Experimental): Covid-19 booster every 6 months and IIV at baseline
  Interventions: Biological: Inactivated influenza vaccine (IIV) at baseline; Biological: COVID-19 Vaccines at a 6-month interval
- Group 4 (Experimental): Covid-19 booster every 6 months and IIV at 1 month
  Interventions: Biological: Inactivated influenza vaccine at Month 1; Biological: COVID-19 Vaccines at a 6-month interval

INTERVENTIONS:
Biological: Inactivated influenza vaccine (IIV) at baseline — National Advisory Committee on Immunization (NACI) recommended seasonal inactivated influenza vaccine for moderate to severely immunocompromised patients by age at baseline
  Arms: Group 1; Group 3
Biological: COVID-19 Vaccines at a 3-month interval — Updated NACI recommended COVID-19 booster for moderate to severely immunocompromised patients at a 3-month interval
  Arms: Group 1; Group 2
Biological: Inactivated influenza vaccine at Month 1 — National Advisory Committee on Immunization (NACI) recommended seasonal inactivated influenza vaccine for moderate to severely immunocompromised patients by age 1-month following initial COVID-19 booster
  Arms: Group 2; Group 4
Biological: COVID-19 Vaccines at a 6-month interval — Updated NACI recommended COVID-19 booster for moderate to severely immunocompromised patients at a 6-month interval
  Arms: Group 3; Group 4

SUMMARY:
The goal of this pragmatic embedded open-label, 2 x 2 factorial phase II randomized controlled trial is to evaluate strategies to improve COVID-19 booster and influenza vaccine immunogenicity in people living with immunocompromising conditions (PLIC).

The main questions it aims to answer are:

1. Is co-administration of seasonal inactivated influenza vaccine (IIV) with the most up-to-date recommended COVID-19 booster dose non-inferior in inducing a 1-month peak protective humoral response against COVID-19, compared to a strategy of sequential administration of COVID-19 booster dose followed by seasonal IIV given one month later?
2. Is the administration of the most up-to-date recommended COVID-19 booster doses at 3-month intervals superior at maintaining a longer term protective humoral immune response, compared to booster doses administered at 6-month intervals?

Researchers will compare (1) COVID-19 and Influenza vaccines administered at Day 0 + COVID-19 Booster at a 3-month interval, (2) COVID-19 vaccine administered at Day 0 and Influenza vaccine administered at Day 28 + COVID-19 Booster at a 3-month interval, (3) COVID-19 and Influenza vaccines administered at Day 0 + COVID-19 Booster at a 6-month interval, and (4) COVID-19 vaccine administered at Day 0 and Influenza vaccine administered at Day 28 + COVID-19 Booster at a 6-month interval to see if median neutralization capacity of patient sera is non-inferior in the co- vs. sequential administration arms at 1-month after the initial COVID-19 booster and superior in the 3-month interval arms vs. the 6-month interval arms at 12 months after the initial COVID-19 booster. These outcomes will also be compared at 2-months for question 1 and 6-months for question 2.

People living with immunocompromising conditions who take part in the trial will have blood samples drawn to verify immune response, be monitored for changes in clinical events and therapies, and complete questionnaires to verify adverse effects, quality of life and economic impact.

DETAILED DESCRIPTION:
Background:

People living with immunocompromising conditions (PLIC) are more susceptible to complications related to respiratory infections. According to Statistics Canada data, in 2020 approximately 14% of Canadians aged 15 years or older suffered from a compromised immune system. PLIC (e.g., solid organ transplant (SOT) recipients, people living with human immunodeficiency viruses (PLWH), inflammatory bowel disease (IBD), or systemic autoimmune rheumatic diseases (RD) are at risk for experiencing a wide range of respiratory infections. A recent North American study assessed the socioeconomic burden associated with immunocompromising conditions. MarketScan datasets from 2017-2021 showed that PLIC accounted for 32% of hospitalizations for acute respiratory infections (representing a 5-8-fold higher risk than in non-immunocompromised hosts).

PLIC are at elevated risk of severe infection and death from COVID-19 increasing burden to patients and healthcare systems. Often including members of diverse ethnocultural origin, PLIC have also been among the most significantly affected by the COVID-19 pandemic. Vaccination is the most effective way to reduce the severity respiratory disease and infection-associated complications in the general population. Yet, suboptimal immune status results in a higher risk for COVID-19-related hospitalization (up to 13-fold) and death (up to 19-fold) compared with the general population in many PLIC, with substantial implications for healthcare burden and costs, despite PLIC comprising but a minority of the overall population.

Immunogenicity and protection from severe disease can be improved in PLIC with COVID-19 booster doses. A systematic review by the COVID-19 evidence network found that PLIC were more susceptible to severe infections and hospitalizations with emerging variants when compared with the general public. This was attributed to immunomodulatory agents (e.g., calcineurin inhibitors, antimetabolites, steroids, cytotoxic therapy, biological response modifiers) impairing the formation of memory T cells, decreasing cellular-mediated immune responses, and limiting capacity to seroconvert and sustain protective immune memory responses. For example, a meta-analysis in SOT found seroconversion and cellular response rates of 39.2% (95% confidence interval [CI], 33.3%-45.3%) and 41.6% (95% CI, 30.0%-53.6%), respectively, after the primary series in solid organ transplant (SOT).

As the pandemic progressed, it was observed that three or four doses of COVID-19 vaccines increased immunogenicity and protected against severe disease requiring hospitalization, with antibody response being most pronounced in the presence of hybrid immunity, arising when SARS-CoV-2 infection was paired with multiple vaccinations. Importantly, decreased immunogenicity has been observed in PLIC in relation to other vaccines, such as the Inactivated Influenza Vaccine (IIV), warranting high-dose (HD) IIV administration to accomplish seroconversion.

Rationale:

The increased risk of COVID-19 and influenza, alongside adverse outcomes of respiratory infections in PLIC and the variability in vaccine responses highlight the need for optimizing immunogenicity and elucidating the mechanisms underlying blunted and/or less durable vaccine responses in PLIC.

Correlates of protective humoral immunity and COVID-19 disease severity. Antigen-binding antibodies, as well as neutralizing antibodies, have been proposed as independent correlates of protection from SARS-CoV-2 infections. The WHO expert committee consensus defined anti-SARS-CoV-2-S1-Receptor-Binding Domain IgG of BAU/mL as low concentrations, 200-300 BAU/mL as mid-range concentrations, and 700-800 BAU/mL as high concentrations. PLIC demonstrated a reduced capacity to mount protective antibody responses. Yet, additional doses resulted in higher antibody concentrations. A recent analysis by De Serres and team demonstrated antibody levels in the range of 700-1200 BAU/ml conferred protection as measured by a surrogate virus neutralization test (sVNT) threshold of 30% against Omicron. Taken together, this body of evidence suggests that neutralizing or binding anti-S could serve as correlates for protection. Importantly, humoral correlates of protection need to also be evaluated for emerging viral variants especially those which have acquired immune-evasion properties. Moreover, in addition to humoral immunity, spike-specific CD4+ and CD8+ T cells are also critical for vaccine-induced protection and are active contributors to global correlates of protection in many individuals.

Correlates of protective cellular immunity. The identification of correlates of cellular immunity capable of informing clinical care has been hampered by a paucity of rapid antigen-specific cellular immunity assays alongside increased costs and time demands. Activation-induced marker (AIM) assays, wherein antigen-specific T cell subsets are enumerated in peripheral blood mononuclear cells (PBMC) identified by their upregulation of AIM (e.g., CD40L, 4-1BB, CD69), are effective at quantifying virus antigen-reactive T cells. However, the rarity of these cells seldom conveys the quality and functional fate of antigen-specific T cell subsets contributing to the global cellular response. Whether AIM phenotypes could be implemented as rapid assays of cellular immunity and exploited towards clinical decision-making, warrants further study.

The trial will provide evidence to guide health policy in a highly diverse and vulnerable subpopulations of PLIC. More specifically, the trial will inform the preferred vaccine schedule for COVID-19 and IIV in these patients, potentially improving upon vaccine acceptance, adherence, and protection, eventually improving burden to patients, caretakers, and the health care system.

Primary Objective(s):

1. To assess whether co-administration of seasonal inactivated influenza vaccine (IIV) with the most up-to-date recommended COVID-19 booster dose is non-inferior in inducing a 1-month peak protective humoral response against COVID-19, compared to a strategy of sequential administration of COVID-19 booster dose followed by seasonal IIV given one month later

   It is hypothesized that the co-administration strategy will be non-inferior to the sequential strategy in inducing a peak 1-month SARS-CoV-2-specific neutralizing antibody response in PLIC. It will also be less costly, with no increase in adverse effects, and no detrimental effect on response to seasonal IIV as measured by hemagglutination inhibition.
2. To assess whether the administration of the most up-to-date recommended COVID-19 booster doses at 3-month intervals is superior at maintaining a longer term protective humoral immune response, compared to booster doses administered at 6-month intervals

It is hypothesized that the 3-month booster strategy will be superior to the 6-month strategy in inducing a SARS-CoV-2--specific neutralizing antibody response that is sustained for 12 months without increasing adverse effects or disease-specific complications.

ELIGIBILITY:
Inclusion Criteria:

- All participants must meet ALL the following inclusion criteria: i. Adults (≥18 years) ii. Received the primary mRNA COVID-19 vaccine series (i.e., ≥3 doses) iii. Have at least one of the following immunocompromising conditions:

a) Received a solid organ transplant (SOT) ≥3-months ago, and treated with a conventional maintenance immunosuppression regimen; b) People living with HIV (PLWH) receiving ART for ≥6 months who meet at least one of the following conditions: i) AIDS-defining illness in the last 6 months, ii) TB diagnosis in the last 6-months, iii) CD4<200 cells/µL in the last 6 months, iv) CD4%<15% in the last 6 months, or v) absence of HIV viral suppression in the last 6 months; c) Inflammatory bowel disease (IBD) treated with a conventional or biologic immunosuppressive agent for ≥3 months; d) Rheumatoid arthritis or systemic lupus erythematosus (herein referred to as rheumatological disease (RD)) treated with a conventional or biologic immunosuppressive agent for ≥3 months.

Exclusion Criteria:

* Potential participants who meet ANY of the following criteria will be excluded:

  i. Received any of the following:
  1. Annual vaccination against influenza < 6 months ago
  2. COVID-19 booster < 3 months ago ii. History of any of the following:

  <!-- -->

  1. life-threatening reaction any component of the IIV or COVID-19 vaccines
  2. Guillain-Barre syndrome or myocarditis within 6 weeks of a previous influenza or COVID-19 vaccination
  3. Contraindication to intramuscular vaccines such as bleeding disorder, severe thrombocytopenia, etc; iii. Receiving intravenous immunoglobulins; iv. Have underlying primary inborn errors of immunity; v. Receiving chemotherapy such as cyclophosphamide < 6-months ago; vi. Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Median neutralization capacity against prevalent SARS-CoV-2 variant | At 1-month and 2-months following the initial COVID-19 booster dose for primary objective 1 and at 12-months and 6-months following initial COVID-19 booster dose for primary objective 2
  Median neutralization capacity of patient sera/plasma from each group, as measured by half maximal inhibitory dilution (ID50) against the prevalent SARS-CoV-2 variant circulating at time of measurement. For objective 1, this outcome will be compared between the co- vs. sequential administration arms at 1-month (T1) after the COVID-19 booster (peak humoral response). This outcome will also be compared at 2-months (T2). For objective 2, this outcome will be compared 12-months (T12) after the first COVID-19 booster between participants who have received COVID-19 boosters at 0, 3, 6 and 9 months (3-month interval arm) vs. those who received COVID-19 booster doses at 0 and 6-months (6-month interval arm). This outcome will also be compared at 6-months (T6).

SECONDARY OUTCOMES:
Median neutralization capacity against ancestral and SARS-CoV-2 variant in vaccine | For primary objective 1, at 1-month and 2-months after the COVID-19 booster. For primary objective 2, at 6 and 12 months
  D50 against the SARS-CoV-2 variant included in the vaccine with measurements against the ancestral variant serving as a reference
Anti-Spike and anti-Nucleocapsid concentrations | Baseline, 1, 2, 4, 6, 7, 10, and 12 months after the first study COVID-19 booster
  Concentration of anti-Spike (response to vaccines) and anti-Nucleocapsid (SARS-CoV-2 infection)
IgA, and IgM antibody concentration | Baseline, 1, 2, 4, 6, 7, 10, and 12 months after the first study COVID-19 booster
  IgA, and IgM antibody concentration against SARS-CoV-2 and IgG1 to 4 subtypes (in a subset of participants)
Hemagglutination inhibition (HI) response | 1 month after IIV
  Hemagglutination inhibition (HI) response for each influenza strain in the vaccine
T-cell responses to SARS-CoV-2 and cytokines assays | Baseline, 1, 2, 4, 6, 7, 10, and 12 months after the first study COVID-19 booster
  T-cell responses to SARS-CoV-2 and cytokine assays (in a subset of participants)
Repeated measures of ID50 | Baseline, 1- and 2-months for objective 1; 4-, 7-, and 10-months for objective 2
  Repeated measures of ID50 against the prevalent, included in the vaccine, and ancestral SARS-CoV-2 variants

OTHER OUTCOMES:
Adverse reactions to the vaccines | Following COVID-19 booster and/or IIV at baseline, 1, 3, 6 and 9-months
  Adverse reactions to the vaccines will be verified by monitoring participants for a period of 30 mins following vaccine administration. Also, self-reported adverse events (Reactogenicity) and their severity will be recorded by patients using a diary for a period of 1-week following each vaccine administration.
Evidence of immune activation | Quarterly (at baseline, 3, 6, 9, and 12-months)
  Evidence of immune activation (e.g., rheumatological or inflammatory bowel disease flares, allograft rejection, or development of donor-specific antibodies)
SARS-CoV-2 infections | Every visit (at baseline, 1, 2, 3, 4, 6, 7, 9, 10, and 12-months)
  Evidence of SARS-CoV-2 infections
Influenza infections | Every visit (at baseline, 1, 2, 3, 4, 6, 7, 9, 10, and 12-months)
  Evidence of Influenza infections
Emergency room visits | Every visit (at baseline, 1, 2, 3, 4, 6, 7, 9, 10, and 12-months)
  Documented emergency room visits
Hospitalizations | Every visit (at baseline, 1, 2, 3, 4, 6, 7, 9, 10, and 12-months)
  Documented hospitalizations
Death | Every visit (at baseline, 1, 2, 3, 4, 6, 7, 9, 10, and 12-months)
  Documented deaths

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes